CLINICAL TRIAL: NCT06640621
Title: A Randomized Controlled Study on the Effect of Brachial Plexus Block with Different Concentrations of Ropivacaine on Diaphragm Movement
Brief Title: The Effect of Brachial Plexus Block on Diaphragm Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M2021684; LM2022383 (Other: Peking University Third Hospital Ethics Commitee)
Record Dates: First submitted 2022-11-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-06

CONDITIONS: Phrenic Paralysis; Shoulder Joint Surgery; Rotator Cuff Injury
Keywords: brachial plexus block; diaphragm movement
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Brachial Plexus Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I (Active Comparator): In group I(high concentration group), ropivacaine 100mg + normal saline to 20ml (0.5% ropivacaine 20ml) is used for single brachial plexus block under ultrasound guidance before general anesthesia.
  Interventions: Drug: Different concentration of ropivacaine for single brachial plexus block
- group II (Experimental): In group II (low concentration group), ropivacaine 40mg + normal saline to 20ml (0.2% ropivacaine 20ml) is used for single brachial plexus block under ultrasound guidance before general anesthesia.
  Interventions: Drug: Different concentration of ropivacaine for single brachial plexus block

INTERVENTIONS:
Drug: Different concentration of ropivacaine for single brachial plexus block — 40 ASA grade I - II patients were selected from the patients who underwent shoulder ligament rupture repair surgery under selective general anesthesia combined with brachial plexus block analgesia in the sports medical center of our hospital. They were randomly divided into two groups: high concentration group (group I) and low concentration group (Group II), with 20 cases in each group. 40 patients underwent a single brachial plexus block under ultrasound guidance before general anesthesia.

SUMMARY:
The purpose of this study is to quickly evaluate the degree of phrenic nerve block by observing the changes of diaphragm movement through ultrasound, and to find the best scheme for clinical application by controlling the concentration of narcotic drugs, so as to reduce respiratory related complications.

DETAILED DESCRIPTION:
40 ASA grade I - II patients were selected from the patients who underwent shoulder ligament rupture repair surgery under selective general anesthesia combined with brachial plexus block analgesia in the sports medical center of our hospital. They were randomly divided into two groups: high concentration group (group I) and low concentration group (Group II), with 20 cases in each group. 40 patients underwent a single brachial plexus block under ultrasound guidance before general anesthesia. In group I, ropivacaine 100mg + normal saline to 20ml (0.5% ropivacaine 20ml), and in group II, ropivacaine 40mg + normal saline to 20ml (0.2% ropivacaine 20ml). The high-frequency ultrasonic probe was located in the intermuscular sulcus, clearly exposing the three trunks of the brachial plexus. Using out of plane technology, the drug solution was injected around the brachial plexus, Ultrasonic images showed that the drug solution evenly wrapped the nerve trunks. The diaphragmatic movement of patients was scanned and recorded before and 30 minutes after block. The dispensing nurse, the operator and the follow-up doctor are independent individuals, and the operator and the follow-up doctor do not know the patient grouping. After confirming the effect of nerve block, the operating doctor will carry out general anesthesia and start the operation. The patients were followed up 6 hours after operation, and NRS scores were made and recorded.

ELIGIBILITY:
Inclusion Criteria:

* operation type: patients undergoing shoulder ligament rupture repair under selective general anesthesia combined with nerve block analgesia
* age: 18 ~ 65
* ASA class I or II

Exclusion Criteria:

* patient rejection
* brachial plexus injury
* severe cardiovascular disease
* allergic to the drugs used in the test
* infection at the puncture site
* difficulty in understanding (unable to understand the pain assessment method)
* recent history of opioid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
the maximum range of motion of bilateral diaphragm | The ultrasound examination of bilateral diaphragms was carried out before brachial plexus block on the affected side, and the ultrasound examination of diaphragm on the blocked side was carried out again 10 minutes after local anesthetic
  Using a low-frequency probe (3-5mhz), place the probe at the bilateral axillary front or at the junction of the clavicular midline and the costal margin respectively, and take the liver and spleen as the sound window, it can be seen that the diaphragm is in an arc-shaped strong echo line. Select the M-mode, and make the sampling line vertical to the diaphragm. Measure the motion amplitude / movement of the diaphragm during calm breathing and maximum deep breathing, and the vertical motion distance (CM) of the diaphragm in the inspiratory phase and expiratory phase respectively.
the change rate of diaphragm thickness | The ultrasound examination of bilateral diaphragms was carried out before brachial plexus block on the affected side, and the ultrasound examination of diaphragm on the blocked side was carried out again 10 minutes after local anesthetic injection
  Select the M-mode to make the sampling line vertical to the diaphragm, Measure the end inspiratory and end expiratory diaphragm thickness at calm breathing and maximum deep breathing respectively, and calculate the change rate of diaphragm thickness at calm breathing and maximum deep breathing [(end inspiratory diaphragm thickness - end expiratory diaphragm thickness) / end expiratory diaphragm thickness × 100%].

SECONDARY OUTCOMES:
Pain relief score of patients. | 6 hours and 24 hours after operation
  NRS score of patients at 6 hours and 24 hours after operation. The Numeric Rating Scale (NRS) is a tool used to assess pain by asking patients to select a number on a scale of 0 to 10 to indicate their level of pain. 0 is painless, 10 is severe .

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No